CLINICAL TRIAL: NCT03190642
Title: Prospective Evaluation of Perioperative Steroid Dosing on Postsurgical Edema in Orthognathic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jean Charles Doucet (Other)
Collaborators: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Jean Charles Doucet, Principal Investigator, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OMFSTEROIDS
Record Dates: First submitted 2017-06-11; First posted 2017-06-19 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Post-operative Edema; Steroid Use
Keywords: Orthognathic Surgery; Swelling
MeSH Terms: interventions — Methylprednisolone; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1000mg methylprednisolone group (Active Comparator): Evaluating effects of 1000mg of methylpresdnisolone administered immediately preoperatively and its effects on swelling.
  Interventions: Drug: Methylprednisolone
- 125mg methylprednisolone group (Active Comparator): Evaluating effects of 125mg of methylpresdnisolone administered immediately preoperatively and its effects on swelling.
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone — Administration of 1000mg vs 125mg methylprednisolone preoperatively in orthognathic surgery.
  Other Names: Solumedrol

SUMMARY:
The current standard of care at the Oral and Maxillofacial Department at the CDHA is the use of one gram of methylprednisolone administered intravenously prior to orthognathic surgery. This is largely based on the work of Habal. The administration of one gram of methylprednisolone can be concerning for the anesthesiologist since this is an unusually large dose of steroid in comparison to use in other surgical specialties. As with most medications, the chances of steroid-related complications increase with increasing doses of steroids.

The researchers are proposing a prospective, double-blind randomized control trial to determine if a smaller dose of methylprednisolone (125mg) can be used safely and effectively instead of one gram of methylprednisolone.

DETAILED DESCRIPTION:
Orthognathic surgery is a commonly performed surgery to correct facial functional and esthetic deformities. At the Atlantic Centre of Oral and Maxillofacial Surgery in Halifax, Nova Scotia, over 300 of these surgeries are carried out yearly. Orthognathic surgery is comprised of procedures performed in both the maxilla and mandible which include Lefort 1, bilateral sagittal split and functional (BSSO) and functional genioplasty. Common sequelae after orthognathic surgery include post-operative pain and swelling.

Swelling occurs almost universally to some degree after orthognathic surgery. Steroid therapy has long been advocated for the reduction of post-operative swelling in oro-facial surgeries, as there is good evidence to support its use for this purpose. In 1978, Habal showed that one gram of methylprednisolone administered in a controlled dog model reduced post-operative swelling. He later carried this over to his practice of cosmetic facial surgeries. His studies have laid the much of the ground work for the use of steroid therapy in head and neck surgeries today.

Other studied benefits of steroid use in facial surgery include decreased post-operative pain, trismus, nausea and vomiting as well as decreased length of hospital stays. Complications of steroid use include compromised healing or infection, sleep disturbances, hyperglycemia, avascular necrosis of bone, steroid-related acne and adverse psychiatric effects.

The use of perioperative steroids as a means of swelling control is the current standard of care in the practice of orthognathic surgery. Despite this fact, there is little consensus on the ideal steroid regimen (i.e. type and dosing) to use for surgery. As such, the use of steroids in Oral and Maxillofacial surgical practices are based primarily on surgeon's preference and familiarity with a particular steroid regimen. This is likely due to the weak evidence in published literature in favor of a steroid regimen to mitigate post-operative swelling.

Most literature in favor of particular steroid regimens involves crude or arbitrary measurements of swelling. In 1978, Habal showed that one gram of methylprednisolone administered in a controlled dog model reduced post-operative swelling. This observation was made by a trained observer against a control group who received no steroid. Other studies have had trained observers look at post-operative photographs of patients who had undergone orthognathic surgery to stratify which had "more" or "less" swelling. Another study attempted to quantify the degree of post-operative swelling by measuring the distance between the earlobes under the chin. These authors acknowledged that this could be altered by the facial movements produced during orthognathic surgery and that better means of measurement of facial swelling should be employed in future research.

The current standard of care at the Oral and Maxillofacial Department at the CDHA is the use of one gram of methylprednisolone administered intravenously prior to orthognathic surgery. This is largely based on the work of Habal. The administration of one gram of methylprednisolone can be concerning for the anesthesiologist since this is an unusually large dose of steroid in comparison to use in other surgical specialties. As with most medications, the chances of steroid-related complications increase with increasing doses of steroids.

The researchers are proposing a prospective, double-blind randomized control trial to determine if a smaller dose of methylprednisolone (125mg) can be used safely and effectively instead of one gram of methylprednisolone, which is the current standard of care in our department. One hundred and twenty-five milligrams of methylprednisolone is a readily available dose of steroids and has been shown in several studies to be effective in the reduction of swelling after oral surgeries and other swelling-related conditions. In their systematic literature review of corticosteroid administration in oral and orthognathic surgery, Dan et al. concluded that a preoperative dose of methylprednisolone >85mg results in a significant decrease in post-operative oedema. The researchers hypothesize that there will be little difference between groups with regards to primary study outcome measure of post-operative swelling.

ELIGIBILITY:
Inclusion Criteria:

* All patients age 14 and over undergoing orthognathic surgery at the Atlantic Centre of Oral and Maxillofacial Surgery in Halifax, Nova Scotia will be included in our study. The clinic is located in the Victoria General Hospital in Halifax, Nova Scotia. Orthognathic surgery includes any combination of Lefort 1, Bilateral Sagittal Split Osteotomy (BSSO) and functional genioplasty procedures.

Exclusion Criteria:

* Patients with pertinent medical history that precludes the use of high-dose steroids will be excluded from our study. This includes:

  * Known hypersensitivity to steroids
  * Type 1 diabetic patients who may have a severe elevation of blood sugars with steroid use.
  * Systemic fungal infections
  * Arrested tuberculosis
  * Herpes simplex keratitis
  * Acute psychoses
  * Cushing's syndrome
  * Peptic ulcer disease
  * Pregnant patients and patients with current infections will be excluded Breast feeding mother

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Post-operative edema | Post-operative period- post-op day 1 until braces off or until 100 weeks post-operatively, whichever comes first
  Measurement of post-operative edema using 3D facial scanner

SECONDARY OUTCOMES:
Patient perceived swelling | Post-operative day 2
  Measurement of post-operative patient perceived swelling via survey
Post-operative pain | Post-operative day 2
  Measurement of post-operative pain via survey
Post-operative sleep | Post-operative day 2
  Measurement of post-operative sleep via survey
Post-operative nausea | Post-operative day 2
  Measurement of post-operative nausea via survey
Length of hospital stay | Until discharge from hospital or post-operative day 100, which ever comes first
  Measurement of length of post-operative hospital stay
Rate of post-operative infection | Post-operative period- post-op day 1 until braces off or until 100 weeks post-operatively, which ever comes first
  Measurement of post-operative infections

CONTACTS AND LOCATIONS:
Locations (1):
- QE II Health Sciences Center, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
NO IPD will be shared with researchers outside of the study

REFERENCES:
- [Background] Guernsey LH, DeChamplain RW. Sequelae and complications of the intraoral sagittal osteotomy in the mandibular rami. Oral Surg Oral Med Oral Pathol. 1971 Aug;32(2):176-92. doi: 10.1016/0030-4220(71)90221-0. No abstract available. PMID 5284103
- [Background] Dan AE, Thygesen TH, Pinholt EM. Corticosteroid administration in oral and orthognathic surgery: a systematic review of the literature and meta-analysis. J Oral Maxillofac Surg. 2010 Sep;68(9):2207-20. doi: 10.1016/j.joms.2010.04.019. Epub 2010 Jun 29. PMID 20591548
- [Background] Habal MB, Powell RD. Experimental facial edema: treatment with methylprednisolone. J Surg Res. 1978 May;24(5):353-8. doi: 10.1016/0022-4804(78)90026-4. No abstract available. PMID 651330
- [Background] Habal MB. Prevention of postoperative facial edema with steroids after facial surgery. Aesthetic Plast Surg. 1985;9(2):69-71. doi: 10.1007/BF01570331. PMID 4025052
- [Background] Chegini S, Dhariwal DK. Review of evidence for the use of steroids in orthognathic surgery. Br J Oral Maxillofac Surg. 2012 Mar;50(2):97-101. doi: 10.1016/j.bjoms.2010.11.019. Epub 2011 Feb 12. PMID 21316821
- [Background] Huaman ET, Juvet LM, Nastri A, Denman WT, Kaban LB, Dodson TB. Changing patterns of hospital length of stay after orthognathic surgery. J Oral Maxillofac Surg. 2008 Mar;66(3):492-7. doi: 10.1016/j.joms.2007.08.025. PMID 18280382
- [Background] Poetker DM, Reh DD. A comprehensive review of the adverse effects of systemic corticosteroids. Otolaryngol Clin North Am. 2010 Aug;43(4):753-68. doi: 10.1016/j.otc.2010.04.003. PMID 20599080
- [Background] Precious DS, Hoffman CD, Miller R. Steroid acne after orthognathic surgery. Oral Surg Oral Med Oral Pathol. 1992 Sep;74(3):279-81. doi: 10.1016/0030-4220(92)90058-x. PMID 1407985
- [Background] Galen DM, Beck M, Buchbinder D. Steroid psychosis after orthognathic surgery: a case report. J Oral Maxillofac Surg. 1997 Mar;55(3):294-7. doi: 10.1016/s0278-2391(97)90546-2. No abstract available. PMID 9054921
- [Background] Weber CR, Griffin JM. Evaluation of dexamethasone for reducing postoperative edema and inflammatory response after orthognathic surgery. J Oral Maxillofac Surg. 1994 Jan;52(1):35-9. doi: 10.1016/0278-2391(94)90010-8. PMID 8263640
- [Background] Widar F, Kashani H, Alsen B, Dahlin C, Rasmusson L. The effects of steroids in preventing facial oedema, pain, and neurosensory disturbances after bilateral sagittal split osteotomy: a randomized controlled trial. Int J Oral Maxillofac Surg. 2015 Feb;44(2):252-8. doi: 10.1016/j.ijom.2014.08.002. Epub 2014 Oct 7. PMID 25304755
- [Background] van der Meer WJ, Dijkstra PU, Visser A, Vissink A, Ren Y. Reliability and validity of measurements of facial swelling with a stereophotogrammetry optical three-dimensional scanner. Br J Oral Maxillofac Surg. 2014 Dec;52(10):922-7. doi: 10.1016/j.bjoms.2014.08.019. Epub 2014 Sep 15. PMID 25219776
- [Background] Lubbers HT, Medinger L, Kruse A, Gratz KW, Matthews F. Precision and accuracy of the 3dMD photogrammetric system in craniomaxillofacial application. J Craniofac Surg. 2010 May;21(3):763-7. doi: 10.1097/SCS.0b013e3181d841f7. PMID 20485043
- [Background] Esen E, Tasar F, Akhan O. Determination of the anti-inflammatory effects of methylprednisolone on the sequelae of third molar surgery. J Oral Maxillofac Surg. 1999 Oct;57(10):1201-6; discussion 1206-8. doi: 10.1016/s0278-2391(99)90486-x. PMID 10513866
- [Background] Ichinose M, Sugiura H, Nagase H, Yamaguchi M, Inoue H, Sagara H, Tamaoki J, Tohda Y, Munakata M, Yamauchi K, Ohta K; Japanese Society of Allergology. Japanese guidelines for adult asthma 2017. Allergol Int. 2017 Apr;66(2):163-189. doi: 10.1016/j.alit.2016.12.005. Epub 2017 Feb 11. PMID 28196638